CLINICAL TRIAL: NCT05896891
Title: San Raffaele EoE Biobank: New Horizons From Etiopathogenesis and Physiopathology
Brief Title: San Raffaele EoE Biobank
Acronym: EoEBiobank
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Silvio Danese, Professor, IRCCS San Raffaele
Other Study IDs: EoE Biobank
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Eosinophilic Esophagitis
Keywords: eosinophilic; disorders; translational
MeSH Terms: conditions — Eosinophilic Esophagitis; Disease | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood, saliva and esophageal tissues
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: esophagogastroduodenoscopy (EGD), buccal swab, blood withdrawal — During routine EGD, biopsy, blood and buccal saliva samples will be withdraw and stored at San Raffaele Hospital

SUMMARY:
Eosinophilic Esophagitis (EoE) is a immuno-mediated disease, characterised by a Th-2 food-antigen driven chronic inflammatory response of the esophagus. Main symptoms are dysphagia and food bolus impaction, frequently overlapping with most atypical and general symptoms like heartburn or regurgitation and difficulty to thrive in children. Overall incidence and prevalence of EoE are rapidly increasing. The complete comprehension of pathogenetic and molecular mechanism underlying this complex and relatively new disease is still to be conquered. For this reason, we created this EoE Biobank, in order to collect blood, oral and esophageal tissue samples of proven EoE patients to further exploit new insights of this disease.

DETAILED DESCRIPTION:
Every EoE patient pertaining to the EoE Unit of San Raffaele Hospital in Milan from 1st June 2023 will be enrolled in the EoE Biobank protocol after being adequately informed and after having signed the informed consent during a preliminary visit where also different clinical and demographic variable of each patient will be taken and stored in an anonymus database. Every patient, during the endoscopic examination performed according to clinical practice guideline for his management, will be asked to provide a sample of oral saliva, 5 mL of blood sample (directly withdraw from the previously placed venous catheter) and additional esophageal biopsies from the esophagus, normally performed for the diagnosis or the follow-up of the disease. The collected samples will be stored in Biological Resources Centre (BRC) of the host organization. These sample will later be analyzed "in vitro" in the context of dedicated protocols

ELIGIBILITY:
Inclusion Criteria:

* EoE diagnosis proven histologically with clinical activity
* Age > 16 years

Exclusion Criteria:

* Not signed informed consent
* No definite EoE diagnosis

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Every male or female patient > 16 years pertaining to IRCCS San Raffaele Hospital in Milan
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-09-12 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Molecular characterization of eosinophilic esophagitis | June 1st 2023 to June 1 st 2026
  Transcriptomic, meta-transcriptomic and molecular staining of different biologic tissues of EoE patients

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Hospital, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: No